CLINICAL TRIAL: NCT00687466
Title: Phase 3 Study on the Efficacy of Slow Release Insulin in Cystic Fibrosis Patients With Glucide Intolerance and Clinical Decay
Brief Title: Study on the Efficacy of Slow Release Insulin in Cystic Fibrosis Patients With Glucide Intolerance and Clinical Decay
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione per la ricerca sulla Fibrosi Cistica (Other)
Responsible Party: Laura Minicucci. MD, Genova CF Center Head, Pediatric Department,CF Center Genova, G.Gaslini Institute, Genova, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFC #21/2006; eudraCT number 2005-002135-27; IGG-FC-G-01
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Cystic Fibrosis; Glucose Intolerance
Keywords: Cystic Fibrosis; Glucose Intolerance
MeSH Terms: conditions — Cystic Fibrosis; Glucose Intolerance | interventions — Insulin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Insulin yes
  Interventions: Drug: Insulin
- 2 (No Intervention): Insulin no

INTERVENTIONS:
Drug: Insulin — Insulin Glargine will be administered subcutaneously at the dosage of 0.1 U/Kg/die for three months. In case no hypoglycemic episodes occur during this period, the dosage will be increased to 0.15 U/Kg/die in occasion of the first control (T1) and will be scheduled for other three months. If even during this latter period no cases no hypoglycemic episodes occur, at the second control (T2) the dosage will be increased to the maximum of 0.2/U/Kg/die. It is generally accepted that the final dosage of glargine can be tailored to each patient, but it should be maintained between 0.1 and 0.2 U/Kg/die.
  Glargine should be administered once daily in the morning and always at the same hour.
  Other Names: Lantus
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate whether the anticipated use of glargine in CF patients with glucose intolerance may prevent the worsening of nutritional status and pulmonary function.

DETAILED DESCRIPTION:
Diabetes mellitus may often complicate the cystic fibrosis course, and it is usually preceded by a condition defined as glucose intolerance, during which a significant decay of patient's general conditions is observed. A slow release insulin (glargine) has become available in the market for diabetic patients: its characteristics allow for a single daily dose, and no need of repeated daily monitoring of glycemia.

In this randomized controlled clinical trial we evaluate whether the anticipated use of glargine in CF patients with glucose intolerance may prevent the worsening of nutritional status and pulmonary function.

Eligible patients who will accept to participate to this study will be randomly allocated in the group who will or will not receive glargine as additional supportive therapy. Patients will in any case continue the CF therapy prescribed by their treating physicians and their usual diet. All the patients will be evaluated every three months to assess their nutritional, pulmonary and glycometabolic status. The follow-up will continue until the 18th month after the study entry.

ELIGIBILITY:
Inclusion Criteria:

* Ascertained diagnosis of CF
* Age ≥ 10 years
* Glucide intolerance: 2 pathologic OGTT ( at 120' glucose value: >140 mg% and <200 mg%) at 2-6 months' interval between each other
* At least one of the following conditions:

  * BMI (body mass index) < 10th centile for age and sex (according to Rolland Cachera 1991)
  * Loss of one BMI centile class for age and sex in the last year (according to Rolland Cachera 1991)
  * FEV1 ≤ 80% of predicted
  * FEV1 decrease ≥ 10% in the last year

Exclusion Criteria:

* Specific contraindications for the use of glargine

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Nutritional status evaluated as variations of Z score of BMI | At recruitment time and at +3, +6, +9, +12, +15, +18 months

SECONDARY OUTCOMES:
Glucose tolerance improvement evaluated as improvement of glycometabolic parameter (glycosylated Hb) | At time recruitment and +3,+6,+9+12+15+18 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Minicucci, MD, Principal Investigator — G.Gaslini Institute Pediatric Department CF Center
Locations (6):
- Italy (6):
  - Pediatric Department, General Hospital,CF Center, Cerignola (Foggia)
  - Ospedale Maggiore Policlinico, Adult CF Center, Milan
  - Pediatric Department, Federico II University, Pediatric CF Center, Napoli
  - Pediatric Department G.De Cristina Hospital CF Center, Palermo
  - Bambino Gesù Hospital CF Center, Roma
  - Policlinico Umberto I. CF Center, Roma

REFERENCES:
- [Background] Moran A, Hardin D, Rodman D, Allen HF, Beall RJ, Borowitz D, Brunzell C, Campbell PW 3rd, Chesrown SE, Duchow C, Fink RJ, Fitzsimmons SC, Hamilton N, Hirsch I, Howenstine MS, Klein DJ, Madhun Z, Pencharz PB, Quittner AL, Robbins MK, Schindler T, Schissel K, Schwarzenberg SJ, Stallings VA, Zipf WB, et al. Diagnosis, screening and management of cystic fibrosis related diabetes mellitus: a consensus conference report. Diabetes Res Clin Pract. 1999 Aug;45(1):61-73. doi: 10.1016/s0168-8227(99)00058-3. No abstract available. PMID 10499886
- [Background] Mackie AD, Thornton SJ, Edenborough FP. Cystic fibrosis-related diabetes. Diabet Med. 2003 Jun;20(6):425-36. doi: 10.1046/j.1464-5491.2003.00924.x. PMID 12786675
- [Background] Solomon MP, Wilson DC, Corey M, Kalnins D, Zielenski J, Tsui LC, Pencharz P, Durie P, Sweezey NB. Glucose intolerance in children with cystic fibrosis. J Pediatr. 2003 Feb;142(2):128-32. doi: 10.1067/mpd.2003.5. PMID 12584532
- [Background] Lanng S, Thorsteinsson B, Nerup J, Koch C. Influence of the development of diabetes mellitus on clinical status in patients with cystic fibrosis. Eur J Pediatr. 1992 Sep;151(9):684-7. doi: 10.1007/BF01957574. PMID 1396931
- [Background] Milla CE, Warwick WJ, Moran A. Trends in pulmonary function in patients with cystic fibrosis correlate with the degree of glucose intolerance at baseline. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):891-5. doi: 10.1164/ajrccm.162.3.9904075. PMID 10988101
- [Background] Dobson L, Hattersley AT, Tiley S, Elworthy S, Oades PJ, Sheldon CD. Clinical improvement in cystic fibrosis with early insulin treatment. Arch Dis Child. 2002 Nov;87(5):430-1. doi: 10.1136/adc.87.5.430. No abstract available. PMID 12390923
- [Background] Rafii M, Chapman K, Stewart C, Kelly E, Hanna A, Wilson DC, Tullis E, Pencharz PB. Changes in response to insulin and the effects of varying glucose tolerance on whole-body protein metabolism in patients with cystic fibrosis. Am J Clin Nutr. 2005 Feb;81(2):421-6. doi: 10.1093/ajcn.81.2.421. PMID 15699230
- [Background] Rolon MA, Benali K, Munck A, Navarro J, Clement A, Tubiana-Rufi N, Czernichow P, Polak M. Cystic fibrosis-related diabetes mellitus: clinical impact of prediabetes and effects of insulin therapy. Acta Paediatr. 2001 Aug;90(8):860-7. PMID 11529531
- [Background] Nousia-Arvanitakis S, Galli-Tsinopoulou A, Karamouzis M. Insulin improves clinical status of patients with cystic-fibrosis-related diabetes mellitus. Acta Paediatr. 2001 May;90(5):515-9. PMID 11430710
- [Background] Dobson L, Sheldon CD, Hattersley AT. Conventional measures underestimate glycaemia in cystic fibrosis patients. Diabet Med. 2004 Jul;21(7):691-6. doi: 10.1111/j.1464-5491.2004.01219.x. PMID 15209760
- [Background] Lombardo F, De Luca F, Rosano M, Sferlazzas C, Lucanto C, Arrigo T, Messina MF, Crisafulli G, Wasniewska M, Valenzise M, Cucinotta D. Natural history of glucose tolerance, beta-cell function and peripheral insulin sensitivity in cystic fibrosis patients with fasting euglycemia. Eur J Endocrinol. 2003 Jul;149(1):53-9. doi: 10.1530/eje.0.1490053. PMID 12824866
- [Background] Bizzarri C, Lucidi V, Ciampalini P, Bella S, Russo B, Cappa M. Clinical effects of early treatment with insulin glargine in patients with cystic fibrosis and impaired glucose tolerance. J Endocrinol Invest. 2006 Mar;29(3):RC1-4. doi: 10.1007/BF03345538. PMID 16682829
- [Background] Bismuth E, Laborde K, Taupin P, Velho G, Ribault V, Jennane F, Grasset E, Sermet I, de Blic J, Lenoir G, Robert JJ. Glucose tolerance and insulin secretion, morbidity, and death in patients with cystic fibrosis. J Pediatr. 2008 Apr;152(4):540-5, 545.e1. doi: 10.1016/j.jpeds.2007.09.025. Epub 2007 Nov 26. PMID 18346512